CLINICAL TRIAL: NCT01886417
Title: Electromyography Study of Lip Muscles During Auditory Verbal Hallucinations Without Subvocalization in Patients With Schizophrenia
Brief Title: Auditory Verbal Hallucinations in Schizophrenia
Acronym: HAV
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: GIPSA-LAB (Other)
Responsible Party: Sponsor
Other Study IDs: 0906; 2009-A00248-49 (Registry Identifier: ID RCB)
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Auditory verbal hallucinations (AVHs) are speech perceptions in the absence of a relevant external stimulation. Some accounts of AVHs claim that a deficit in inner speech monitoring would cause the verbal thoughts of the patient to be perceived as external voices resulting in AVHs.

In order to examine whether AVHs correspond to self-generated inner speech, the present study aims at collecting speech muscle activity during covert AVHs (without articulation), overt speech and rest. Surface electromyography (sEMG) is used on schizophrenia patients and control subjects to detect any speech muscle activity during AVH.

ELIGIBILITY:
Inclusion Criteria:

Healthy controls:

* must be more than 18 years and less than 60 years old
* pre-inclusion medical examination
* must have signed consent form
* must be able to read stimuli on a screen

Schizophrenia patients:

* must be more than 18 years and less than 60 years old
* pre-inclusion medical examination
* must have signed consent form
* must be able to read stimuli on a screen
* diagnosed with a schizophrenia disorder according to DSM-IV TR (diagnostic and statistical of mental disorders) (PANSS item P3 greater than 4)
* prior evaluation of the secondary effects of any medication via Barnes and AIMS scales
* affiliated with the French social security
* if under guardianship, must have additional consent form signed by guardian

Exclusion Criteria:

Healthy controls:

* if aged less than 18 years or more than 60 years
* diagnosed with any psychiatric disorder
* with any language disorder (aphasia, SLI, dysarthria, stuttering, etc.)
* with auditory impairment
* pregnant, parturient, breast-feeding

Schizophrenia patients:

* if aged less than 18 years or more than 60 years
* significant secondary effects of antipsychotic medication, measured with the Barnes and AIMS scales
* with a neurodegenerative disease
* with any language disorder (aphasia, SLI, dysarthria, stuttering, etc.)
* with auditory impairment
* pregnant, parturient, breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: in- and out-patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Labial EMG activity during auditory verbal hallucination | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Thierry BOUGEROL, MD, PHD, HDR, Principal Investigator — University Hospital of Grenoble, France
Locations (1):
- University Hospital of Grenoble, Grenoble, France